CLINICAL TRIAL: NCT07161245
Title: A Randomized Clinical Trial on the Improvement of Fatigue in Patients With Primary Biliary Cholangitis by Implementation of a Multimodal Rehabilitation Program and Study of Its Pathophysiological Mechanisms
Brief Title: RELIEF: Multimodal Prehabilitation to Treat Fatigue in Patients With Primary Biliary Cholangitis
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RELIEF/2025
Record Dates: First submitted 2025-06-02; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: FATIGUE; PREHABILITATION; PHYSICAL ACTIVITY; MINDFULNESS MEDITATION; NUTRITION; QUALITY OF LIFE
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fatigue; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants with primary biliary cholangitis (PBC) under follow-up in hepatology outpatient clinics who present with moderate to severe fatigue, as defined by a score greater than 29 on the PBC-40 questionnaire, and who agree to participate in the study after providing informed consent, will be eligible for inclusion.
  Once enrolled, participants with PBC and fatigue will be randomly assigned to either receive the multimodal intervention for 8 weeks or be allocated to the control group. Randomization will be performed using simple randomization via the REDCap platform. For the control group, after the initial 8-week period, the opportunity to participate in the multimodal rehabilitation program will be offered. Subsequently, both groups, after completing the 8-week intervention, will continue with the remote phase of the program for an additional six months of follow-up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal prehabilitation (Experimental): 8 weeks program of tailored physical exercise program with nutritional and psychological counselling to be carried out to a patient on the basis of his/her health condition, social circumstances and adherence profile.
  Interventions: Other: Multimodal prehabilitation
- Standard of care (Other): Standard Counselling: Patients in the control group will follow standard of care of the hospital and will be given general recommendations on physical activity, nutrition and stress/anxiety management.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: Multimodal prehabilitation — The multimodal prehabilitation program will consist of:
  1. twice-weekly supervised exercise training at the hospital gym for approximately 8 weeks (induction phase), followed by 16 weeks of telematic, supervised, home-based exercise (maintenance phase);
  2. nutritional consultation, including diet optimization and supplementation if needed;
  3. individual or group-based psychological support.
  Arms: Multimodal prehabilitation
Other: standard of care — Participants in the control group will follow the standard of care provided by the hospital and will receive general recommendations on physical activity, nutrition, and stress/anxiety management.
  Arms: Standard of care

SUMMARY:
The implementation of a non-pharmacological multimodal intervention program-including physical exercise, nutritional counseling, and psychological support-is expected to improve fatigue in patients with primary biliary cholangitis. Consequently, this improvement is anticipated to enhance quality of life and cognitive symptoms, while also positively impacting emotional, social, and occupational aspects.

From a pathophysiological perspective, it is hypothesized that chronic cholestasis and/or immune system activation, with the release of pro-inflammatory cytokines, leads to both central and peripheral alterations causing fatigue.

At the central level, systemic inflammation may induce neuronal senescence in the basal ganglia, resulting in altered functional connectivity networks dependent on these regions and/or structural and connectivity changes in areas involved in interoception, such as the insula and anterior cingulate cortex.

At the peripheral level, the hypothesis is that chronic inflammation mediated by anti-mitochondrial antibodies causes mitochondrial metabolic dysfunction in muscle cells, which would be reflected in changes observed in the gene expression analysis of these cells.

Improvement in fatigue following the multimodal intervention program is expected to be associated with normalization of the immunological profile, enhanced functional brain connectivity, and improved mitochondrial metabolism in muscle.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is a rare autoimmune disease that damages the small bile ducts and primarily affects women. Although it is a liver disease, its most common symptom is fatigue, affecting up to 60% of patients. Fatigue is a debilitating symptom, described by patients as "a brain fog" that causes concentration problems and memory loss, along with "a lack of energy" that leads to poor exercise tolerance and early exhaustion. This significantly impacts quality of life, negatively affecting family, social, and work-related activities. To the frustration of both patients and healthcare providers, fatigue is not correlated with the severity of liver disease, and there is currently no effective treatment.

Ursodeoxycholic acid (UDCA), the first-line treatment for PBC, has been shown to improve disease survival, but it does not appear to have an effect on fatigue, as demonstrated by a meta-analysis. Other treatments, such as bezafibrate, have also failed to show improvement in fatigue. Several clinical trials have tested treatments targeting different pathophysiological mechanisms, including selective serotonin reuptake inhibitors (SSRIs), stimulants like modafinil, and immunomodulatory therapies such as rituximab, all with negative results.

Currently, new drugs have been approved as second-line treatments for PBC, such as elafibranor and seladelpar. The latter may have some impact on fatigue; however, this was not the primary objective of the study, and the mechanisms associated with this improvement remain unclear.

One of the main reasons why no treatment exists is the lack of understanding of the underlying mechanisms. Fatigue is a complex and likely multifactorial symptom. It has been hypothesized that chronic immune system activation, leading to excessive production of inflammatory substances, could be a trigger. Additionally, it remains unknown whether alterations in bile acid composition, which are molecules with potent biological effects on multiple organs, could worsen fatigue. Furthermore, this chronic inflammation may induce changes in both the brain and muscles, contributing to the development of fatigue.

It has been demonstrated that physical exercise reduces systemic inflammation by lowering inflammatory substances and can also improve abnormalities in muscle energy production. Studies conducted in patients with other diseases associated with fatigue, such as multiple sclerosis, have shown that exercise programs can be beneficial for fatigue management.

At present, experience with physical training programs for PBC patients with fatigue is very limited. The results of a study conducted in the United Kingdom and another in Canada suggest that a home-based exercise program may improve fatigue. However, both studies have certain limitations, as the follow-up was remote, there was no supervision to ensure proper execution of the exercises or that they were performed at the prescribed intensity. Additionally, the effective exercise duration was only about 15 minutes, which, along with its moderate intensity, is unlikely to induce specific adaptations in mitochondrial biogenesis and efficiency. On the other hand, while patients with liver diseases generally express positive attitudes toward the benefits of supervised exercise, they also acknowledge a lack of confidence in initiating it independently.

Based on this evidence, an integrated exercise program is proposed, consisting of two phases: an initial supervised phase lasting eight weeks and a subsequent remote phase, combined with nutritional counseling and psychological support. It is hypothesized that this program will improve fatigue and consequently enhance quality of life, as well as alleviate associated cognitive symptoms (such as depression and sleep disturbances).

To better understand the changes occurring in the organs involved in fatigue, the investigators aim to analyze immune responses and bile acids to determine their potential association with fatigue, as has been observed in other autoimmune diseases. Additionally, potential alterations at both the brain and muscle levels will be explored.

At the neurological level, functional connectivity alterations in brain regions involved in fatigue will be studied using functional magnetic resonance imaging (fMRI). At the muscular level, changes in muscle metabolism will be analyzed by studying gene expression in muscle fibers. Muscle samples will be obtained using a minimally invasive technique called muscle microbiopsy, which involves a fine-needle puncture of a muscle and is not associated with complications. These studies will be conducted before and after the exercise program, aiming to observe the positive changes expected at all levels.

These studies will be conducted before and after the training program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* PBC diagnosis according to EASL guidelines
* Moderate - severe fatigue defined by ≥ 29 points in PBC-40 questionnaire

Exclusion Criteria:

* Age > 80 years
* Severe pruritus
* Decompensated cirrhosis
* Other causes of liver disease than PBC
* Liver transplant (LT) o placement on a waiting-list for LT
* Uncontrolled thyroid disesase
* Anemia with haemoglobin <11g/dl
* Uncontrolled cardiovascular risk factors
* BMI > 35,
* Acute myocardial infarct or unstable angina the past 6 months
* Muscle disease or systemic disease with potential muscle involvement
* Dysautonomy
* Untreated osteoporosis
* Untreated celiac disease
* Alcohol consumption > 14 standard drinks (SD) in women and >21 (SD) in men per week
* Chronic kidney disease ≥ 4 KDIGO stage
* Malignancy in the past two years (except for non melanoma skin cancer and in situ cervical carcinoma)
* Not capable of performing or following the prehabilitation program
* Involvement in a clinical trial the previous 2 months
* Refusal of informed consent

For the study of the pathophysiology of fatigue, additional exclusion criteria will be established: Severe depression or neuropsychiatric disease, 2) Treatment with centrally acting drugs, 3) Muscular or systemic disease with potential muscle involvement, 4) Immunosuppressive treatment, 5) Sleep disorder, 6) Obesity (BMI >30).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Severity Assessed by PBC-40 | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  To evaluate the effect of a non-pharmacological multimodal intervention program on fatigue severity and its impact in participants with primary biliary cholangitis (PBC). Fatigue will be assessed using the Primary Biliary Cholangitis-40 (PBC-40) fatigue domain, which consists of 11 items scored from 1 to 5. Scoring Range: 11 to 55; higher scores indicate greater fatigue.
Change in Fatigue Severity Assessed by Visual Analogue Scale | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  To evaluate the effect of a non-pharmacological multimodal intervention program on fatigue severity and its impact in participants with primary biliary cholangitis (PBC). Fatigue will be assessed using the Visual Analogue Scale (VAS) for fatigue, which captures the participant's perception of fatigue severity. Scoring Range: 0 (no fatigue) to 10 (worst imaginable fatigue).
Change in Fatigue Impact Assessed by Fatigue Impact Scale (FIS) | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  To evaluate the effect of a non-pharmacological multimodal intervention program on fatigue severity and its impact in participants with primary biliary cholangitis (PBC). Fatigue will be assessed using the Modified Fatigue Impact Scale (MFIS), which assesses the impact of fatigue on physical, cognitive, and psychosocial functioning. Scoring Range: 0 to 84; higher scores indicate greater fatigue-related impairment

SECONDARY OUTCOMES:
Change in Cognitive Symptoms Assessed by PBC-40 | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To evaluate changes in cognitive symptoms using the Primary Biliary Cholangitis-40 (PBC-40) questionnaire. The cognitive domain ranges from 6 to 30 points. Higher scores indicate worse symptoms.
Change in Extrahepatic Symptoms Assessed by PBC-40 | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To evaluate changes in extrahepatic symptoms using the Primary Biliary Cholangitis-40 (PBC-40) questionnaire. The symptoms domain ranges from 7 to 35 points. Higher scores indicate worse symptoms.
Change in Quality of Life Assessed by EQ-5D-5L Index Score | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To assess health-related quality of life using only the EQ-5D-5L index score derived from five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The index score ranges from -0.594 to 1, where higher scores indicate better health status.
Change in Self-Perceived Health Status Assessed by EQ Visual Analogue Scale | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To evaluate self-perceived overall health using the EQ Visual Analogue Scale (EQ-VAS), part of the EQ-5D-5L instrument, reported separately. The EQ-VAS ranges from 0 to 100, where 0 = worst imaginable health and 100 = best imaginable health.
Change in Disability Assessed by the WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To measure disability and functional impairment. Scoring Range: 0 to 100; higher scores indicate greater disability.
Change in Anxiety and Depression Assessed by the Hospital Anxiety and Depression Scale (HADS) | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To evaluate levels of anxiety and depression. Scoring Range: 0 to 21 for each subscale (anxiety and depression); higher scores indicate greater symptom severity.
Change in Sleep Quality Assessed by the Epworth Sleepiness Scale (ESS) | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To assess daytime sleepiness as a proxy for sleep quality. Scoring Range: 0 to 24; higher scores indicate greater daytime sleepiness.
Change in Work Productivity and Activity Impairment Assessed by the WPAI Questionnaire | Baseline, week 8 and/or after the exercise phase, and end of trial.
  To measure absenteeism and work productivity impairment. Percentage scores for absenteeism, presenteeism, overall work impairment, and activity impairment; higher percentages indicate greater impairment.
Change in Systemic Inflammation Assessed by Pro-Inflammatory Cytokines | Baseline and end of induction phase (2 months) for participants with fatigue; single time point for control groups.
  To evaluate systemic inflammation and bile acid metabolism by analyzing a panel of pro-inflammatory cytokines (measured via ELISA), lysophosphatidic acid, autotaxin, and bile acids. Each biomarker will be quantified by the laboratory using standardized assays.
  Units of Measure: Concentrations reported in appropriate laboratory units (e.g., pg/mL, nmol/L) depending on the biomarker.
Functional Connectivity Alterations in Brain Regions Assessed by fMRI. | Baseline and end of induction phase (2 months) for participants with fatigue; single time point for control groups.
  To examine changes in functional connectivity in gray matter regions, including the basal ganglia and insula, using functional magnetic resonance imaging (fMRI).
Changes in Muscle Mitochondrial Metabolism Assessed by Gene Expression Analysis | Baseline and end of induction phase (2 months) for participants with fatigue; single time point for control groups.
  To analyze gene expression profiles related to mitochondrial metabolism in muscle fibers obtained via muscle microbiopsy. Units of measure: Relative gene expression (fold change compared to baseline or control).
Change in Aerobic Capacity | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  Aerobic capacity will be evaluated to measure changes in functional exercise tolerance using the 6-Minute Walk Test (6MWT), which measures distance walked in meters (0-700 m typical; higher distances = better capacity).
  Unit of Measure: Meters.
Change in Physical Activity Levels | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  Physical activity levels will be assessed to determine changes in habitual activity, with scores ranging from 0 to 142, where higher scores indicate greater overall physical activity.
Change in Frailty Status | Baseline (week 0), post-intervention (week 8), and end of maintenance phase (6 months).
  Frailty will be evaluated using the Liver Frailty Index (LFI), a continuous scale derived from a combination of grip strength, chair-stand time, and balance testing. In adult liver disease populations, median LFI values range approximately from 2.7 in individuals without liver disease to 3.6 in those with cirrhosis. Established thresholds classify LFI scores of < 3.2 as "robust", 3.2-4.4 as "prefrail", and > 4.4 as "frail"
Feasibility and Satisfaction of a Multimodal Rehabilitation Program for the Treatment of Fatigue | From enrollment to the end of treatment at 6 months
  Participant experience will be assessed using satisfaction questionnaires. Adherence to the intervention and loss to follow-up will be evaluated by analyzing reasons for non-compliance or withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Rodríguez Tajes, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Marta Ubré Lorenzo, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz-Feijoo B, Agusti N, Sebio R, Siso M, Carreras-Dieguez N, Domingo S, Diaz-Cambronero O, Torne A, Martinez-Palli G, Arguis MJ. A multimodal prehabilitation program for the reduction of post-operative complications after surgery in advanced ovarian cancer under an ERAS pathway: a randomized multicenter trial (SOPHIE). Int J Gynecol Cancer. 2022 Nov 7;32(11):1463-1468. doi: 10.1136/ijgc-2022-003652. PMID 35793862
- [Background] Gimeno-Santos E, Coca-Martinez M, Arguis MJ, Navarro R, Lopez-Hernandez A, Castel MA, Romano B, Lopez-Baamonde M, Sandoval E, Farrero M, Sanz M, Bofill A, Martinez-Palli G. Multimodal prehabilitation as a promising strategy for preventing physical deconditioning on the heart transplant waiting list. Eur J Prev Cardiol. 2020 Dec;27(19):2367-2370. doi: 10.1177/2047487319889709. Epub 2019 Nov 25. No abstract available. PMID 31766879
- [Background] Barberan-Garcia A, Ubre M, Pascual-Argente N, Risco R, Faner J, Balust J, Lacy AM, Puig-Junoy J, Roca J, Martinez-Palli G. Post-discharge impact and cost-consequence analysis of prehabilitation in high-risk patients undergoing major abdominal surgery: secondary results from a randomised controlled trial. Br J Anaesth. 2019 Oct;123(4):450-456. doi: 10.1016/j.bja.2019.05.032. Epub 2019 Jun 25. PMID 31248644
- [Background] Williams FR, Vallance A, Faulkner T, Towey J, Kyte D, Durman S, Johnson J, Holt A, Perera MT, Ferguson J, Armstrong MJ. Home-based exercise therapy in patients awaiting liver transplantation: protocol for an observational feasibility trial. BMJ Open. 2018 Jan 21;8(1):e019298. doi: 10.1136/bmjopen-2017-019298. PMID 29358444
- [Background] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811
- [Background] Watt M, Hyde A, Johnson E, Wright GM, Vander Well S, Sadasivan C, Lee-Baggley D, Spence JC, Mason A, Ko HH, Tam E, Tandon P. An online mind-body program improves mental health and quality of life in primary biliary cholangitis: A randomized controlled trial. Hepatol Commun. 2023 Nov 6;7(11):e0316. doi: 10.1097/HC9.0000000000000316. eCollection 2023 Nov 1. PMID 38346279
- [Background] Freer A, Williams FR, Durman S, Hayden J, Armstrong MJ, Trivedi PJ. A home-based exercise programme attenuates fatigue in primary biliary cholangitis: Results from the EXCITED clinical trial. JHEP Rep. 2024 Sep 6;6(12):101210. doi: 10.1016/j.jhepr.2024.101210. eCollection 2024 Dec. PMID 39640219
- [Background] Kowdley KV, Bowlus CL, Levy C, Akarca US, Alvares-da-Silva MR, Andreone P, Arrese M, Corpechot C, Francque SM, Heneghan MA, Invernizzi P, Jones D, Kruger FC, Lawitz E, Mayo MJ, Shiffman ML, Swain MG, Valera JM, Vargas V, Vierling JM, Villamil A, Addy C, Dietrich J, Germain JM, Mazain S, Rafailovic D, Tadde B, Miller B, Shu J, Zein CO, Schattenberg JM; ELATIVE Study Investigators' Group; ELATIVE Study Investigators' Group. Efficacy and Safety of Elafibranor in Primary Biliary Cholangitis. N Engl J Med. 2024 Feb 29;390(9):795-805. doi: 10.1056/NEJMoa2306185. Epub 2023 Nov 13. PMID 37962077
- [Background] Jopson L, Newton JL, Palmer J, Floudas A, Isaacs J, Qian J, Wilkinson J, Trenell M, Blamire A, Howel D, Jones DE. RITPBC: B-cell depleting therapy (rituximab) as a treatment for fatigue in primary biliary cirrhosis: study protocol for a randomised controlled trial. BMJ Open. 2015 Aug 20;5(8):e007985. doi: 10.1136/bmjopen-2015-007985. PMID 26297361
- [Background] Talwalkar JA, Donlinger JJ, Gossard AA, Keach JC, Jorgensen RA, Petz JC, Lindor KD. Fluoxetine for the treatment of fatigue in primary biliary cirrhosis: a randomized, double-blind controlled trial. Dig Dis Sci. 2006 Nov;51(11):1985-91. doi: 10.1007/s10620-006-9397-5. Epub 2006 Oct 20. PMID 17053955
- [Background] Silveira MG, Gossard AA, Stahler AC, Jorgensen RA, Petz JL, Ali AH, Lindor KD. A Randomized, Placebo-Controlled Clinical Trial of Efficacy and Safety: Modafinil in the Treatment of Fatigue in Patients With Primary Biliary Cirrhosis. Am J Ther. 2017 Mar/Apr;24(2):e167-e176. doi: 10.1097/MJT.0000000000000387. PMID 27148676
- [Background] Lee JY, Danford CJ, Trivedi HD, Tapper EB, Patwardhan VR, Bonder A. Treatment of Fatigue in Primary Biliary Cholangitis: A Systematic Review and Meta-Analysis. Dig Dis Sci. 2019 Aug;64(8):2338-2350. doi: 10.1007/s10620-019-5457-5. Epub 2019 Jan 10. PMID 30632051
- [Background] Hollingsworth KG, Newton JL, Taylor R, McDonald C, Palmer JM, Blamire AM, Jones DE. Pilot study of peripheral muscle function in primary biliary cirrhosis: potential implications for fatigue pathogenesis. Clin Gastroenterol Hepatol. 2008 Sep;6(9):1041-8. doi: 10.1016/j.cgh.2008.04.013. Epub 2008 Aug 8. PMID 18691944
- [Background] Yeaman SJ, Kirby JA, Jones DE. Autoreactive responses to pyruvate dehydrogenase complex in the pathogenesis of primary biliary cirrhosis. Immunol Rev. 2000 Apr;174:238-49. doi: 10.1034/j.1600-0528.2002.00021h.x. PMID 10807520
- [Background] Hollingsworth KG, Newton JL, Robinson L, Taylor R, Blamire AM, Jones DE. Loss of capacity to recover from acidosis in repeat exercise is strongly associated with fatigue in primary biliary cirrhosis. J Hepatol. 2010 Jul;53(1):155-61. doi: 10.1016/j.jhep.2010.02.022. Epub 2010 Mar 31. PMID 20447719
- [Background] Goldblatt J, James OF, Jones DE. Grip strength and subjective fatigue in patients with primary biliary cirrhosis. JAMA. 2001 May 2;285(17):2196-7. doi: 10.1001/jama.285.17.2196. No abstract available. PMID 11325320
- [Background] Mosher VAL, Swain MG, Pang JXQ, Kaplan GG, Sharkey KA, MacQueen GM, Goodyear BG. Primary Biliary Cholangitis Alters Functional Connections of the Brain's Deep Gray Matter. Clin Transl Gastroenterol. 2017 Jul 27;8(7):e107. doi: 10.1038/ctg.2017.34. PMID 28749455
- [Background] D'Mello C, Swain MG. Liver-brain interactions in inflammatory liver diseases: implications for fatigue and mood disorders. Brain Behav Immun. 2014 Jan;35:9-20. doi: 10.1016/j.bbi.2013.10.009. Epub 2013 Oct 16. PMID 24140301
- [Background] Capuron L, Pagnoni G, Drake DF, Woolwine BJ, Spivey JR, Crowe RJ, Votaw JR, Goodman MM, Miller AH. Dopaminergic mechanisms of reduced basal ganglia responses to hedonic reward during interferon alfa administration. Arch Gen Psychiatry. 2012 Oct;69(10):1044-53. doi: 10.1001/archgenpsychiatry.2011.2094. PMID 23026954
- [Background] Dantzer R, Heijnen CJ, Kavelaars A, Laye S, Capuron L. The neuroimmune basis of fatigue. Trends Neurosci. 2014 Jan;37(1):39-46. doi: 10.1016/j.tins.2013.10.003. Epub 2013 Nov 13. PMID 24239063
- [Background] Nelson T, Zhang LX, Guo H, Nacul L, Song X. Brainstem Abnormalities in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Scoping Review and Evaluation of Magnetic Resonance Imaging Findings. Front Neurol. 2021 Dec 17;12:769511. doi: 10.3389/fneur.2021.769511. eCollection 2021. PMID 34975729
- [Background] Zeng J, Fan J, Zhou H. Bile acid-mediated signaling in cholestatic liver diseases. Cell Biosci. 2023 Apr 29;13(1):77. doi: 10.1186/s13578-023-01035-1. PMID 37120573
- [Background] Ronca V, Davies SP, Oo YH, Lleo A. The immunological landscape of primary biliary cholangitis: Mechanisms and therapeutic prospects. Hepatology. 2025 Oct 1;82(4):877-894. doi: 10.1097/HEP.0000000000001225. Epub 2025 Jan 3. PMID 39774114
- [Background] Borren NZ, van der Woude CJ, Ananthakrishnan AN. Fatigue in IBD: epidemiology, pathophysiology and management. Nat Rev Gastroenterol Hepatol. 2019 Apr;16(4):247-259. doi: 10.1038/s41575-018-0091-9. PMID 30531816
- [Background] Jopson L, Jones DE. Fatigue in Primary Biliary Cirrhosis: Prevalence, Pathogenesis and Management. Dig Dis. 2015;33 Suppl 2:109-14. doi: 10.1159/000440757. Epub 2015 Dec 7. PMID 26641884
- [Background] Ismond KP, Aziz B, Wright GM, Mason AL. Self-reported experiences of patients living with primary biliary cholangitis (PBC): Are we treating the liver but not the patient? Can Liver J. 2019 Feb 25;2(1):45-47. doi: 10.3138/canlivj.2018-0017. eCollection 2019 Winter. No abstract available. PMID 35991832
- [Background] Lynch EN, Campani C, Innocenti T, Dragoni G, Biagini MR, Forte P, Galli A. Understanding fatigue in primary biliary cholangitis: From pathophysiology to treatment perspectives. World J Hepatol. 2022 Jun 27;14(6):1111-1119. doi: 10.4254/wjh.v14.i6.1111. PMID 35978669
- [Background] Bjornsson E, Kalaitzakis E, Neuhauser M, Enders F, Maetzel H, Chapman RW, Talwalkar J, Lindor K, Jorgensen R. Fatigue measurements in patients with primary biliary cirrhosis and the risk of mortality during follow-up. Liver Int. 2010 Feb;30(2):251-8. doi: 10.1111/j.1478-3231.2009.02160.x. Epub 2009 Nov 17. PMID 19922590
- [Background] Wunsch E, Stadnik A, Kruk B, Szczepankiewicz B, Kotarska K, Krawczyk M, Gornicka B, Wojcicki M, Milkiewicz P. Chronic Fatigue Persists in a Significant Proportion of Female Patients After Transplantation for Primary Sclerosing Cholangitis. Liver Transpl. 2021 Jul;27(7):1032-1040. doi: 10.1002/lt.26033. Epub 2021 Apr 21. PMID 33641247
- [Background] Jacoby A, Rannard A, Buck D, Bhala N, Newton JL, James OF, Jones DE. Development, validation, and evaluation of the PBC-40, a disease specific health related quality of life measure for primary biliary cirrhosis. Gut. 2005 Nov;54(11):1622-9. doi: 10.1136/gut.2005.065862. Epub 2005 Jun 16. PMID 15961522
- [Background] Montali L, Gragnano A, Miglioretti M, Frigerio A, Vecchio L, Gerussi A, Cristoferi L, Ronca V, D'Amato D, O'Donnell SE, Mancuso C, Luca M, Yagi M, Reig A, Jopson L, Pilar S, Jones D, Pares A, Mells G, Tanaka A, Carbone M, Invernizzi P. Quality of life in patients with primary biliary cholangitis: A cross-geographical comparison. J Transl Autoimmun. 2021 Jan 6;4:100081. doi: 10.1016/j.jtauto.2021.100081. eCollection 2021. PMID 33554101
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: The diagnosis and management of patients with primary biliary cholangitis. J Hepatol. 2017 Jul;67(1):145-172. doi: 10.1016/j.jhep.2017.03.022. Epub 2017 Apr 18. PMID 28427765